CLINICAL TRIAL: NCT02395159
Title: Reduction of Groin Wound Infections After Vascular Surgery in Patients With Risk Factors by the Use a Negative Pressure Wound Incision Management System (KCI Prevena)
Brief Title: Reduction of Groin Wound Infections After Vascular Surgery by Using an Incision Management System (IMS)
Acronym: IMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-048
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Infections
Keywords: vascular surgery patients; wound management
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevena™ IMS (Experimental): The patients in the experimental arm will be treated with the Prevena™ IMS seven days after the surgery
  Interventions: Device: Prevena™ IMS
- sterile plaster dressings (Other): The wound will be treated with the conventional wound management method of sterile plaster dressing.
  Interventions: Other: sterile plaster dressings

INTERVENTIONS:
Device: Prevena™ IMS — Prevena™ IMS is intended for the management of the surgical incision environment and surrounding healthy skin in patients with a risk of postoperative complications such as infections. This entails the maintenance of a closed environment around the incision by applying a negative pressure wound therapy system.
  The corresponding dressing is known under the name Prevena™ Dressing. The layer closest to the skin comprises silver foil, which reduces the microbial colonisation of cells.
  Arms: Prevena™ IMS
Other: sterile plaster dressings — standard wound management method of sterile plaster dressings
  Arms: sterile plaster dressings

SUMMARY:
Comparison of the Prevena™ IMS with the standard wound management method of sterile plaster in vascular surgery patients.

DETAILED DESCRIPTION:
Comparison of the Prevena™ IMS with the standard wound management method of sterile plaster in vascular surgery patients.

The aim is to demonstrate that the application of the Prevena™ IMS significantly reduces the incidence of postoperative wound infections. The wound infections will be classified according to Szilagyi.

The treatment phase begins following vascular surgery with wound management using either the Prevena™ IMS or a standard wound dressing, depending on the group to which the patient was randomly assigned. It involves a minimum stay of 7 and maximum 10 days in hospital.

ELIGIBILITY:
Inclusion Criteria:

* vascular surgery via right or left inguinal approach
* nicotine abuse (active or according to medical condition)
* risk factors:

  1. cardiac risk factors (arterial hypertension, coronary heart disease, status after myocardial infarction)
  2. metabolic disorders (diabetes mellitus type I type II, lipopathy or hyperhomocysteinemia) or chronic or acute renal insufficiency
* previous vascular surgery with inguinal approach
* signed informed consent form
* persons who are legally competent and mentally able to comprehend and follow the instructions of study personnel

Exclusion Criteria:

* local skin infections (fungal infections, acne)
* pregnant and breast-feeding women
* simultaneous participation in another clinical trial
* persons who have been committed to an institution by court or administrative order
* persons in a dependency or employment relationship with the sponsor or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
wound infections | 7 days after the surgery
  The primary objective is the occurrence of inguinal wound infections following surgery. Wound infections will be classified according to Szilagyi.

SECONDARY OUTCOMES:
length of hospital stay | up to 10 days
antibiotic therapy | up to 30 days
revision surgery | up to 30 days
necessity of alternative wound dressings | up to 30 days
prolongation of ambulant treatment | up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Grommes, Principal Investigator — University Hospital, Aachen
Locations (2):
- Germany (2):
  - University Hospital Aachen, vascular surgery, Aachen
  - Marienhospital Wiiten, vascular surgery, Witten

REFERENCES:
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- [Derived] Cristino MA, Nakano LC, Vasconcelos V, Correia RM, Flumignan RL. Prevention of infection in aortic or aortoiliac peripheral arterial reconstruction. Cochrane Database Syst Rev. 2025 Apr 22;4(4):CD015192. doi: 10.1002/14651858.CD015192.pub2. PMID 40260835